CLINICAL TRIAL: NCT03444883
Title: A Multicenter, Randomized, Parallel, Double Blind, Placebo-controlled Phase III Study to Evaluate Safety and Efficacy of Ilaprazole 20mg in Patients With Non-erosive Reflux Disease(NERD)
Brief Title: Phase III Study to Evaluate Safety and Efficacy of Ilaprazole in Patients With NERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IL49NE03
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Non-erosive Reflux Disease
Keywords: NERD; PPI; Ilaprazole
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — ilaprazole

STUDY DESIGN:
Intervention Model Description: A mulicenter, randomized, parallel, double blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): 10mg Ilaprazole x 2 tablets
  Interventions: Drug: Ilaprazole
- Control Group (Placebo Comparator): 10mg placebo of Ilaprazole x 2 tablets
  Interventions: Drug: Ilaprazole

INTERVENTIONS:
Drug: Ilaprazole — 10mgx2 tablet once daily for weeks
  Other Names: IY81149

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ilaprazole 20 mg in patients with non-erosive reflux disease. This study intends to demonstrate the clinical superiority of Ilaprazole 20 mg to placebo administered once daily for 4 weeks.

DETAILED DESCRIPTION:
This study is multicenter, randomized, parallel, double blind, placebo-controlled phase III study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 19 years and ≤ 80 years
2. Diagnosed with non-erosive reflux disease meeting all of the following criteria:

   2-1) At least either heartburn or acid regurgitation has persisted for at least past 3 months before screening 2-2) Have experienced at least either heartburn or acid regurgitation of moderate or higher intensity on at least 2 days of 7 days prior to initiation of the investigational product 2-3) Esophageal mucosal breaks by LA Classification are not observed on upper gastrointestinal endoscopy at screening
3. Voluntarily provide written informed consent to participate in this study

Exclusion Criteria:

1. Esophageal stenosis, ulcerative stenosis, esophagogastric varices or Barrett esophagus confirmed by past upper gastrointestinal endoscopy within 1 year prior to screening
2. Active peptic ulcer or gastrointestinal bleeding confirmed by past upper gastrointestinal endoscopy at screening or within 4 weeks prior to screening
3. Abnormal value on laboratory test at screening:

   3-1) Total Bilirubin, Creatinine > Upper limit of normal (ULN) x 1.5 3-2) Alkaline Phosphatase, BUN > ULN x 2
4. Clinically significant abnormal findings on ECG (major arrhythmia, multifocal PVC, second-degree or higher AV block, etc.) within 3 months prior to screening
5. Have taken H2 receptor antagonists (H2RA), prostaglandin preparations, mucosal protective drugs, prokinetics, etc. within 2 weeks prior to initiation of the investigational product administration, or has taken PPIs within 4 weeks prior to initiation of the investigational product administration
6. Expected to continuously take nonsteroidal antiinflammatory drugs (NSAIDs) including aspirin or steroid preparations during the study
7. Surgical or medical condition that may significantly influence the absorption, distribution, metabolism or excretion of drug, including but not limited to: history of major gastrointestinal surgery such as gastrectomy, gastroenterostomy, colectomy, gastric bypass, gastric ligation or gastric banding; presence or history of active inflammatory bowel disease within 12 months prior to screening; has undergone critical surgery that may influence gastric acid secretion with exception of surgeries such as appendectomy, cholecystectomy, and hysterectomy
8. Zollinger-Ellison syndrome; past history of alcoholism or drug abuse
9. Past history of allergic symptoms (rash, fever, pruritus, etc.) or hypersensitivity to any ingredient of the Investigational product
10. Past history of treated or untreated malignancy, with or without local recurrence or metastasis, within 5 years prior to screening (with exception of local basal cell carcinoma of skin)
11. Pregnant or nursing women
12. Women of childbearing potential who do not use proper contraception during the study
13. Active liver disease; ALT or AST > ULN x 2 at screening; or history of hepatic encephalopathy, esophageal varix, or portacaval shunt
14. Receiving renal dialysis or history of kidney transplantation or presence of severe renal impairment (stage 4 or 5 chronic renal disease)
15. Participated in another clinical study and took an investigational product within 3 months prior to screening
16. Considered by the investigator to be ineligible to participate in this study for other reasons

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Rate of loss of esophagitis symptom at 4 weeks of treatment vs pre-dose | 4 weeks(28 days)
  Percentage of subjects who were assessed as having 'lost' the frequency and intensity of typical esophagitis symptoms by RDQ assessment at 4 weeks of treatment

SECONDARY OUTCOMES:
Chang in esophagitis symptom score at 4 weeks of treatment vs pre-dose | 4 weeks(28 days)
  The mean scores for esophagitis symptom (heartburn and/or acid regurgitation) frequency and intensity assessed with RDQ (Questions a, b/c, d) and the change in mean score across both domains.
Change in PAGI-QoL score at 4 weeks of treatment vs pre-dose | 4 weeks(28 days)
  The change in mean score for quality of life assessed with PAGI-QoL
Change in esophagitis symptom score according to the maximum number of rescue medication doses per day | 4 weeks(28 days)
  The mean scores for esophagitis symptom (heartburn and/or acid regurgitation) frequency and intensity assessed with RDQ (Questions a, b/c, d) at 4 weeks of treatment versus pre-dose according to the maximum number of rescue medication doses per day and the change in mean score across both domains.

CONTACTS AND LOCATIONS:
Overall Officials: DongHo Lee, MD.PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (11):
- South Korea (11):
  - Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu
  - Inje University Busan Paik Hospital, Busan, Busanjin-gu
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Dongjak-gu
  - Chonbuk National University Hospital, Jeonju, Jeonju-si
  - Kangbuk Samsung Hospital, Sungkyunkwan University, Seoul, Jongno-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Inje University Seoul Paik Hospital, Seoul, Jung-gu
  - Severance Hospital Yonsei University Health System, Seoul, Seodaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu
  - Soon Chun Hyang University Hospital, Buchon, Bucheon-si, Wonmi-gu
  - Ewha Womans University Mokdong Hospital, Seoul, Yangcheon-gu

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to other researchers.